CLINICAL TRIAL: NCT03290222
Title: Translation, Adaptation Into Portuguese (Brazilian Culture) and Validation of the Test for Respiratory and Asthma Control in Kids (TRACK)
Brief Title: TRACK: Validation of the Portuguese Version
Acronym: TRACK
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Gustavo Wandalsen, Professor of the Pediatrics Department, Federal University of São Paulo
Other Study IDs: ESR-16-12088
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Asthma; Respiratory Disease
Keywords: Respiratory symptoms; Children
MeSH Terms: conditions — Asthma; Respiration Disorders; Signs and Symptoms, Respiratory

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TRACK: Children will be followed for four weeks (3 to 5 weeks) after the inclusion in the study. Parents will complete the TRACK questionnaire in both visit and will answer additional questions about respiratory symptoms and use of medication.
  Interventions: Other: TRACK questionnaire

INTERVENTIONS:
Other: TRACK questionnaire — TRACK questionnaire consists of five questions, scored 0-20, to be made to caregivers of children with asthma or recurrent respiratory symptoms, regarding respiratory symptoms, nocturnal awakenings and limitation of daily activities in the last four weeks, use of bronchodilators in the last three months and systemic corticosteroids in the last year

SUMMARY:
The TRACK ("Test for Respiratory and Asthma Control in Kids") questionnaire is a validated instrument to evaluate the control of respiratory symptoms in young children. The TRACK questionnaire was developed in English and a version in Portuguese is not available or validated, purpose of the present project.

DETAILED DESCRIPTION:
The TRACK ("Test for Respiratory and Asthma Control in Kids") questionnaire is the only instrument developed and validated so far to evaluate the control of respiratory symptoms in young children under five years of age. The TRACK questionnaire consists of five questions, scored from 0 to 20, given to caregivers of children with asthma or recurrent respiratory symptoms, and addresses respiratory symptoms, nocturnal awakenings and limitation of daily activities in the last four weeks, use of bronchodilator medications over the past three months and systemic corticosteroids in the last year.

The TRACK questionnaire was developed in English and has already been translated and validated into Spanish and Arabic. At the moment there is no translation and validation of the TRACK questionnaire for the Portuguese language, purpose of the present project.

ELIGIBILITY:
Inclusion Criteria:

* Native Portuguese speakers families
* Medical diagnosis of asthma or history of at least three episodes of cough and/or wheeze and/or dyspnea (duration longer than 24 hours) and treated with bronchodilators

Exclusion Criteria:

* Other relevant pulmonary diseases (i.e.: cystic fibrosis, bronchopulmonary dysplasia)
* Systemic diseases (i.e.: heart diseases, neurologic disorders)
* Premature birth (under 37 weeks of gestational age)
* Congenital malformations
* Illiteracy and/or inability of parents to understand the questionnaire

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children up to five years of age with recurrent respiratory symptoms attended at pediatric clinics will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Global Initiative for Asthma (GINA) criteria | 4 weeks
  The TRACK criterion validation will be performed by the comparison of the scores obtained from patients in the three levels of control, according to GINA criteria
Respiratory symptoms | 4 weeks
  Constructive validation will be done by comparing the TRACK notes between patients discriminated according to their respiratory symptoms (symptomatic, recent symptoms, and asymptomatic)

SECONDARY OUTCOMES:
Medical opinion | 4 weeks
  Constructive validation will also be done by comparing the TRACK notes between patients discriminated according to the medical opinion

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Allergy and Clinical Immunology, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murphy KR, Zeiger RS, Kosinski M, Chipps B, Mellon M, Schatz M, Lampl K, Hanlon JT, Ramachandran S. Test for respiratory and asthma control in kids (TRACK): a caregiver-completed questionnaire for preschool-aged children. J Allergy Clin Immunol. 2009 Apr;123(4):833-9.e9. doi: 10.1016/j.jaci.2009.01.058. PMID 19348922
- [Background] Zeiger RS, Mellon M, Chipps B, Murphy KR, Schatz M, Kosinski M, Lampl K, Ramachandran S. Test for Respiratory and Asthma Control in Kids (TRACK): clinically meaningful changes in score. J Allergy Clin Immunol. 2011 Nov;128(5):983-8. doi: 10.1016/j.jaci.2011.08.010. Epub 2011 Sep 8. PMID 21906790
- [Background] Rodriguez-Martinez CE, Nino G, Castro-Rodriguez JA. Validation of the Spanish version of the Test for Respiratory and Asthma Control in Kids (TRACK) in a population of Hispanic preschoolers. J Allergy Clin Immunol Pract. 2014 May-Jun;2(3):326-31.e3. doi: 10.1016/j.jaip.2014.01.014. Epub 2014 Mar 29. PMID 24811025
- [Derived] Wandalsen GF, Dias RG, Chong-Neto HJ, Rosario N, Moraes L, Wandalsen NF, Medeiros D, Bianca ACD, Urrutia-Pereira M, Avila J, Jorge PP, Sole D. Test for Respiratory and Asthma Control in Kids (TRACK): validation of the Portuguese version. World Allergy Organ J. 2018 Dec 5;11(1):40. doi: 10.1186/s40413-018-0219-y. eCollection 2018. PMID 30534341